CLINICAL TRIAL: NCT06345391
Title: The Added Value of Pain Science Education for Children Living Beyond Cancer (PANACEA): Co-creation
Brief Title: Co-creation of Pain Science Education for Children Living Beyond Cancer
Acronym: PANACEA
Status: Not yet recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); University Ghent (Other); University Hospital, Ghent (Other); University of Calgary (Other)
Responsible Party: Principal Investigator, Emma Rheel, PhD, Principal Investigator, Vrije Universiteit Brussel
Other Study IDs: PANACEA_CO-CREATION_2024
Record Dates: First submitted 2024-03-15; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Children Living Beyond Cancer (i.e. Child Cancer Survivor)
Keywords: children living beyond cancer; pain science education; co-creation; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children living beyond cancer: Children between 8-12 years with a history of any cancer diagnosis that are currently in the early survivorship phase (<2y post-treatment).
  Interventions: Other: Co-creation
- Parents of children living beyond cancer: Parents of children (8-12 years) living beyond cancer.
  Interventions: Other: Co-creation
- Pediatric oncology clinicians: Clinicians (e.g. physician, nurse, physical therapist, occupational therapist, psychologist, child life specialist) currently employed in pediatric oncology.
  Interventions: Other: Concept Mapping

INTERVENTIONS:
Other: Co-creation — Participatory approach maximally and directly involving important stakeholders (bottom-up) to co-create a pain science education intervention for children living beyond cancer.
  Groups: Children living beyond cancer; Parents of children living beyond cancer
Other: Concept Mapping — Concept mapping to create a pain science education intervention for children living beyond cancer.
  Groups: Pediatric oncology clinicians

SUMMARY:
A pain science education (PSE) intervention for children (8-12y) living beyond cancer (CBC) will be developed through a co-creational approach with CBC, their parents and pediatric oncology clinicians. The study will be guided by the Intervention Mapping Protocol.

DETAILED DESCRIPTION:
PARTICIPANT RECRUITMENT STRATEGY

Co-creation is a bottom-up approach directly involving the end-users in developing the intervention. For the co-creation of the PSE intervention, 3 groups will be formed: children (8-12yo) living beyond cancer (CBC), their parents, and pediatric oncology clinicians. For each group, 6 to 8 participants will be recruited.

Using purposeful sampling, CBC and their parents will be recruited through various ways, including through patient lists of the participating hospitals (University Hospital Brussels and University Hospital Ghent), by convenience sampling (e.g. research team's networks, social media calls), and through snowball sampling (i.e. participating child-parent dyads encourage other dyads). Taking into account the cognitive and emotional development of children, the age range of CBC is set at 8-12y to restrain wide variation in developmental stage.

Pediatric oncology clinicians (e.g., physicians, physiotherapists, nurses, psychologists, child life specialists, occupational therapists) will be recruited from the participating hospitals and through the research team's networks.

CBC, their parents, and pediatric oncology clinicians can only be included in the study if they meet the inclusion criteria and after written informed consent is obtained. All CBC, parents, and pediatric oncology clinicians will receive verbal and written information on all aspects of the study prior to consent for participation. CBC wishing to participate without a parent will not be excluded, but will still require parental consent.

SAMPLE SIZE CALCULATION

A recent report of the Belgium Cancer Registry stated that annually 360 children between 0-18y are diagnosed with cancer, of which about 90 children of 8-12y. According to the Belgian Cancer Registry the 5-year survival rate for this age group is about 93%, resulting in an estimated 83 CBC per year that can be recruited for the current study. Hence, the foreseen recruitment rate of 6 to 8 participants seems feasible.

RISK MANAGEMENT

In case of slow recruitment of CBC and their parents, additional recruitment sources will be contacted to participate and share the recruitment flyers. In case of slow recruitment of oncology clinicians, other Flemish University hospitals will be approached through the research team's networks.

BASELINE ASSESSMENT

One week before the first session clinical and socio-demographic characteristics of participating CBC, parents and pediatric oncology clinicians will be assessed through a battery of online questionnaires. Questionnaires will be completed using REDCap, a secure web platform for building and managing online databases and surveys (↑ study feasibility, ↑ data protection). The following socio-demographic and clinical information will be collected:

CBC (parent-reported): age, sex, diagnosis date and description, cancer treatment(s) received, treating hospitals, other medical history, current or previous pain treatments (psychosocial, physical, and/or pharmacological).

Parents: age, gender identification, family situation, education level, occupation, and health status.

Oncology clinicians: age, gender, occupation, hospital where they are working, work experience in pediatric oncology, experience with pain education, health status.

CO-CREATION SESSIONS AND CONCEPT MAPPING SESSIONS

For the development of the PSE intervention, 6 co-creation sessions will be organized with CBC and their parents separately, and 3 sessions using concept mapping will be organized with pediatric oncology clinicians.

The co-creation and concept mapping sessions will be guided by the Intervention Mapping Protocol (IMP). The IMP is being used worldwide as the standard protocol for the development, implementation, and evaluation of health promoting interventions.

The content of the co-creation sessions with CBC and their parents will be as follows:

Session 1: explanation of the study aim, assessment of the needs, barriers and facilitators for behavioral change and the outcome expectations of the PSE intervention

Session 2-3: determination of performance objectives and change objectives of the PSE intervention

Session 4-5: selection of practical strategies (content, format, delivery method, timing, materials)

Session 6: demonstration of the co-created PSE intervention, followed by a discussion and evaluation of the developed PSE intervention in terms of satisfaction, understandability, empowerment, and ownership.

The concept mapping sessions with pediatric oncology clinicians will be structured as follows:

Session 1: participants will be asked to answer one key question covering the scope and intention of the study: 'How would you approach a pain science education intervention for CBC?' Answers will be collected through a 'round circle principle'.

Session 2: a card sorting task will be given to the participants in which they are asked to sort the answers of the previous concept mapping session by theme into different piles. After completing the card sorting task, they will have to rate each theme in terms of relevance (population-level effect), modifiability, and expected outcomes on a scale from 1 to 10. With this input, we will proceed to the co-creation sessions with CBC living beyond cancer and their parents.

Session 3: after the co-creation sessions with CBC and their parents, when the PSE intervention becomes more concrete, final feedback on the co-created PSE intervention will be requested from the pediatric oncology clinicians who are willing to be part of the advisory committee.

Results of the co-creation sessions and concept mapping sessions will be cross-validated after each session to end up with one final PSE intervention. Each session will be audio-taped after assent/consent from the participants, to ensure that no valuable information regarding the intervention development process will be lost. All audiotapes will be transcribed and will not be used for any other study purposes. The audiotapes will be deleted after study completion.

PAIN SCIENCE EDUCATION

Pain science education (PSE) is a non-pharmacological pain management approach that aims to facilitate one's understanding of pain mechanisms. It provides a foundation for other pain management strategies by addressing conceptual gaps and misconceptions regarding pain, and by decreasing the perceived threat value of pain.

In terms of the content of the PSE intervention, an interdisciplinary expert panel identified 7 target concepts to form the foundation of a PSE curriculum for children: 1) pain is a protector; 2) the pain system can become overprotective; 3) pain is a brain output; 4) pain is not an accurate marker of tissue stage; 5) there are many potential contributors to one's pain; 6) we are all bioplastic and; 7) pain education is treatment. These 7 success ingredients of PSE will be presented, yet will be open for discussion and will be supplemented with cancer-specific target concepts. Hence, the concrete PSE intervention for CBC will be developed during the co-creation process, so the PSE intervention will not yet be applied/implemented.

ELIGIBILITY:
Inclusion Criteria:

Children living beyond cancer:

* history of (any) cancer diagnosis
* age 8-12y at the time of inclusion
* <2y post-treatment completion (early survivorship phase)
* fluently Dutch speaking and reading
* having access to internet/computer (in order to complete online questionnaires)
* signed informed consent form

Parents of children living beyond cancer:

* fluently Dutch speaking and reading
* having access to internet/computer (in order to complete online questionnaires)
* signed informed consent form

Pediatric oncology clinicians:

* currently employed as a physician, nurse, physical therapist, occupational therapist, psychologist, or child life specialist in pediatric oncology
* fluently Dutch speaking and reading
* having access to internet/computer (in order to complete online questionnaires)

Exclusion Criteria:

Children living beyond cancer:

• presence of psychiatric disorders or severe intellectual disability

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children living beyond cancer and their parents will be recruited through patients lists of the participating hospitals (i.e. University Hospital Brussels and University Hospital Ghent), by convenience sampling (e.g. through the research team's networks, calls on social media), and through snowball sampling (i.e. participating dyads search for and encourage other dyads to participate). Oncology clinicians will be recruited from the participating hospitals by email invitation and through the research team's networks. All eligible children, parents, and oncology clinicians will be informed about the study and receive a consent form.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the co-created intervention | at the end of the last co-creation/concept mapping session, approximately 6 months
  Information about satisfaction of stakeholders (i.e. children living beyond cancer, their parents, and pediatric oncology clinicians) with various aspects of the co-created PSE intervention (e.g., content, complexity, comfort, delivery, and credibility) will be assessed through a small self-developed questionnaire at the end of the last co-creation and concept mapping session. The items of the questionnaire will be based on the ultimately developed intervention and will also include an open-ended question assessing to what extent the developed PSE intervention is what they needed, with the opportunity to suggest alternative treatment content.

SECONDARY OUTCOMES:
Understandability of the co-created intervention | at the end of the last co-creation/concept mapping session, approximately 6 months
  Information about understandability of stakeholders (i.e. children living beyond cancer, their parents, and pediatric oncology clinicians) with regard to the developed PSE intervention through a small self-developed questionnaire.
Empowerment with regard to the co-created intervention | at the end of the last co-creation/concept mapping session, approximately 6 months
  Information about empowerment (self-efficacy, self-esteem, perceived stress and social support) of stakeholders (i.e. children living beyond cancer, their parents, and pediatric oncology clinicians) with various aspects of the co-created PSE intervention will be assessed through a small self-developed questionnaire at the end of the last co-creation and concept mapping session.
Ownership of the intervention development | at the end of each co-creation/concept mapping session, up to 6 months
  Information about ownership (i.e. retention rates throughout the sessions) of stakeholders (i.e. children living beyond cancer, their parents, and pediatric oncology clinicians) will be assessed through a logbook.

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Jette, Brussels Capital, Belgium